CLINICAL TRIAL: NCT06661577
Title: A Multi-Centre Observational Study For The Collection Of A Raman Spectral Database Using The LumAssure Device In Adult Participants Undergoing Dermatological Assessment Of Skin Conditions
Brief Title: An Observational Study Using The LumAssure Device In Participants Undergoing Assessment Of Skin Conditions.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Auckland UniServices Ltd. (Industry); Counties Manukau Health (Other)
Responsible Party: Principal Investigator, Michel Nieuwoudt, Senior Research Fellow, Principal Investigator, The School of Chemical Sciences, University of Auckland, New Zealand
Other Study IDs: HDEC21297; HDEC 21297 (Other: New Zealand Health and Disabilities Ethics Committee)
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Skin Cancers - Basal Cell Carcinoma; Skin Cancers - Squamous Cell Carcinoma; Melanoma of Skin; Inflammatory Dermatoses; Acral Melanoma; Benign Skin Nevus; Benign Skin Tumor
Keywords: skin cancers; melanoma; diagnostic device
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Nevus; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Male and female healthy volunteers, aged 18 years or over, attending a study specific skin check appointment, without a diagnosis or histology of malignancies.
- SOC Patients: Participants attending a standard of care medical appointment at a skin clinic, a plastic surgery or a general practitioner for assessment, diagnosis and/or potential excision of a skin condition, With confirmatory medical practitioner diagnosis, and where appropriate confirmatory histological analysis of excised tissues

SUMMARY:
This is an observational study in adult males and females utilising skin condition measurements using the LumAssure Raman device. Data will be used to determine accuracy under the ROC curve (AUCROC) of the LumAssure device for differentiating between benign and cancerous skin conditions. The measurements will provide data which will be used to establish spectral parameters for different skin conditions. Measurements will be benchmarked against diagnoses from medical specialists, and when available confirmed with histological data.

The main question it aims to answer is :

What is the accuracy, in terms of the area under the ROC curve (AUCROC) of the LumAssure device for differentiating between benign skin conditions and skin cancers in adult males and females? Participants include males and females aged ≥18 years who are undergoing assessment of a skin condition (a lesion or rash) by a dermatologist, general practitioner, or plastic surgeon. Participants' attending the clinics will have their skin conditions examined by a clinician. The LumAssure device will then be used to measure Raman spectra of skin conditions and marked by the clinician. The Raman measurements will be benchmarked against skin condition assessment and, where available, diagnosis by a dermatologist, general practitioner, or a plastic surgeon, and for those lesions undergoing biopsy, confirmed with histology data.

DETAILED DESCRIPTION:
For this observational study, Raman spectra will be measured in the clinic using the LumAssure device, on patients attending standard of care medical clinics (SOC participants) for skin assessments and/or biopsies, and on healthy volunteers attending a clinical research centre (HV participants). The LumAssure device was developed and utilised in a previous proof of concept study (https://doi.org/10.1016/j.xjidi.2023.100238). Development of a robust classification algorithm capable of distinguishing between malignant vs benign skin conditions requires the collection of clinical measurements from a large and diverse participant population with varied skin Fitzpatrick types.

Participants will be recruited via advertising. All participants must provide informed consent prior to study participation and data collection. SOC participants lesions of interest will be identified for LumAssure measurement by their medical specialist during their clinical visit.

Participant data will be de-identified, utilizing a unique study number, and entered directly into an electronic data capture system.

The study will be conducted in accordance with the protocol and applicable regulatory requirements. Participant rights and safety, and study data integrity will be monitored by an independent contract research organization in accordance with the protocol and established procedures.

Approximately 1,600 - 3,000 skin conditions assessment data point cases required from an estimated 400-750 participants (with an estimated 1-4 lesions per participant) will be collected for this study. The participant sample size has been determined by an independent biostatistician. The Protocol established criteria for data handling, management and analysis in order to achieve the primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Male or female aged 18 years or over.
* Willing to undergo a LumAssure device measurement on at least 1 skin condition
* (For Standard of Care patients): are undergoing a skin examination and/or tissue excision by a qualified specialist
* (For Healthy volunteers): are attending a skin check at a study clinic

Exclusion Criteria:

* Tattoo on the skin condition to be measured
* Skin conditions on or directly around the eye area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first group of participants (healthy volunteers), will be those who can attend a free skin check at the Clinical Research Centre at the University of Auckland medical school. The second group of participants (patients referred to/attending a clinic for a skin assessment) will be those attending one of five clinics in the city of Auckland and towns of Dargaville and Hokianga, in New Zealand.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-12-13 (Estimated); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Sufficient numbers of measurements to achieve an acceptable area under the ROC curve (AUCROC) for accurate differentiation between benign skin conditions and skin cancers | Day 1, baseline, 12 months
  The primary endpoint of the study will be the area under the ROC curve (AUCROC) of the LumAssure Raman device measurements for the differentiation between benign skin conditions and skin cancers. The primary aim is to collect sufficient LumAssure Raman device measurements of skin conditions to develop an algorithm which can help detect diagnosed skin conditions and malignancies determined via histological analysis of biopsied samples.

SECONDARY OUTCOMES:
Number of participants with adverse events and descriptions of adverse events | Day 1, baseline, 12 months
  Secondary endpoints:
  The number of participants with adverse events will be recorded, and the types of adverse events will be describes and categorized according to severity (high, medium or low risk).

OTHER OUTCOMES:
Number and type of device inadequacies | Day1, baseline, 12 months
  Recording of the number and types of issues encountered with device function or performance, and categorized according to low, medium or high risk.

CONTACTS AND LOCATIONS:
Overall Officials: Michel K Nieuwoudt, PhD, Principal Investigator — The University of Auckland
Locations (2):
- New Zealand (2):
  - Manukau Super clinic, Auckland
  - Sir Willliam Manchester Plastic surgery suite, Middlemore Hosptial, Auckland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in a publication on the study will be made available. This includes information about the demographics, age, sex, Skin Fitzpatrick type and history of skin cancer of individual participants, which will be de-identified and compiled with the corresponding Raman spectral data into a dataset for data analysis for publication on the study. This dataset can be made available in a data repository upon reasonable request, as is required by many journals for publication.
Supporting Information: CSR
Time Frame: 6 months after completion of the observational study
Access Criteria: Report will be put into a web repository